CLINICAL TRIAL: NCT02527876
Title: Exercise to Promote Quit Attempts in Young Adults
Brief Title: Exercise, Activity and Smoking in Young Adults
Acronym: EASY-A
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Researcher left University
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1505m70321
Record Dates: First submitted 2015-08-05; First posted 2015-08-19 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Exercise, Delayed Control
Keywords: Exercise; Smoking
MeSH Terms: conditions — Motor Activity; Smoking | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Intensity Interval Training/FitBit Flex (Experimental): Meet with personal trainer once per week for 20-minute exercise session
  Interventions: Behavioral: High Intensity Interval Training; Device: FitBit Flex
- Moderate Intensity/FitBit Flex (Experimental): Meet with personal trainer once per week for 30-minute exercise session and exercise two times a week outside of personal trainer
  Interventions: Behavioral: Moderate Intensity; Device: FitBit Flex
- Delayed Control/FtBit Flex (Placebo Comparator): No exercise offered
  Interventions: Behavioral: Delayed Control; Device: FitBit Flex

INTERVENTIONS:
Behavioral: High Intensity Interval Training — High Intensity Interval Training
  Other Names: FitBit Flex
  Arms: High Intensity Interval Training/FitBit Flex
Behavioral: Moderate Intensity — Moderate Intensity Training
  Arms: Moderate Intensity/FitBit Flex
Behavioral: Delayed Control — Delayed Control
  Arms: Delayed Control/FtBit Flex
Device: FitBit Flex — Use to measure increase in Physical Activity

SUMMARY:
The purpose of this study is to evaluate how physical activity levels change in young adults when they start a specific exercise program.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate how physical activity levels change in young adults when they start a specific exercise program. Physical activity levels will be monitored daily via a FitBit Flex. Outcome measures include number of minutes of activity per day and distance traveled per day.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old,
* stable physical/mental health,
* current smoker
* currently minimally active,
* ambulatory,
* interested in increasing their physical activity,
* willingness to attend weekly exercise intervention sessions at a SNAP Fitness location within 10 miles of the University of Minnesota campus,
* the ability to comply with the study protocol and provide informed consent

Exclusion Criteria:

* Contraindications to increasing physical activity including, but not limited to,
* abnormal electrocardiogram or V02 test results,
* high blood pressure (defined as systolic blood pressure over 165 or diastolic blood pressure over 100),
* heart attack, acute (2 days) cardiac event or stroke in preceding six months,
* unstable angina,
* uncontrolled dysrhythmias causing hemodynamic compromise,
* symptomatic severe aortic stenosis,
* uncontrolled symptomatic heart failure,
* acute pulmonary embolism or pulmonary infarction,
* acute myocarditis or
* pericarditis,
* dissecting aneurism,
* acute systemic infection and
* unstable pulmonary or cardiovascular conditions.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Increase in Physical Activity as assessed by FitBit | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Allen, PhD, Principal Investigator — University of Minnesota
Locations (1):
- DCRU, Minneapolis, Minnesota, United States